CLINICAL TRIAL: NCT03022760
Title: Return to Work Among Patients With Stress Related Mental Disorders - An Intervention in the Swedish Primary Care (PRIMA)
Brief Title: Return to Work Among Patients With Stress Related Mental Disorders - An Intervention in the Swedish Primary Care
Acronym: PRIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISM 03-2015
Record Dates: First submitted 2016-11-01; First posted 2017-01-16 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Stress, Psychological; Burnout, Professional; Adjustment Disorders
Keywords: Exhaustion Disorder
MeSH Terms: conditions — Stress, Psychological; Burnout, Professional; Adjustment Disorders

ARMS (2):
- Work-related measures (Active Comparator): * One-day training for GP:s and rehabilitation coordinators
  * A treatment protocol which includes contact with the patient's employer
  * Clinical support from the Institute of Stress Medicine
  Interventions: Behavioral: Work-related measures
- Treatment as usual (No Intervention)

INTERVENTIONS:
Behavioral: Work-related measures — After mapping the patient's psychosocial work situation using tools provided at the one-day training, the patient's employer will be contacted and involved in the rehabilitation planning.
  Arms: Work-related measures

SUMMARY:
The aim of this project is to develop a model for return to work (RTW) for patients sick listed due to stress related mental disorders, which takes into account each patient's specific situation; includes the workplace, and is well adapted to the Swedish primary care setting.

In late 2016, general practitioners (GPs) and rehabilitation coordinators at both public and private primary care centers will be offered a one-day training about work and workability for patients with stress related mental disorders. Also, the participants will be trained in a specific method that includes the patient's employer early in the rehabilitation process

The project has a quasi-experimental and longitudinal design. The intervention will be conducted on 15 different primary care centers, which will be matched with a comparison group. Return to work for 500 patients will be analyzed using registry data, 6, 12 and 18 months after sick-listing. The hypothesis is that patients who are sick-listed at primary care centers that completely or partially implemented the specific method on average will return earlier to work than patients sick-listed at primary care centers that did not implement the method.

Alongside studying if the intervention has an effect on the patients' RTW over time, the investigators aim to investigate the mechanisms explaining the effects and the individual and organizational level (primary care units) circumstances necessary for these mechanisms to be triggered. To gain deeper knowledge about mechanisms and context, the investigators will conduct interviews with the treatment staff and collect registry data about the primary care units.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of International Classification of Diseases (ICD)10 F43
* Has an employment
* Good command in spoken and written Swedish

Exclusion Criteria:

* Participants must not have been on long term sick-leave (>60 days) during the last three years, regardless of causative diagnosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Following sick leave data from the Swedish Social Insurance Agency's records we will measure time taken to return to work (RTW) among patients in the intervention group vs. time taken to RTW among patients in the control group. | Three measurement time points. First measurement will occur 6 months from baseline.
Following sick leave data from the Swedish Social Insurance Agency's records we will measure time taken to return to work (RTW) among patients in the intervention group vs. time taken to RTW among patients in the control group. | Second measurement time point will occur at 12 months from baseline.
Following sick leave data from the Swedish Social Insurance Agency's records we will measure time taken to return to work (RTW) among patients in the intervention group vs. time taken to RTW among patients in the control group. | Third measurement time point will occur at 18 months from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Björk, Study Director — the Institute of Stress Medicine
Locations (1):
- Gothenburg, Sweden

REFERENCES:
- [Derived] Beno A, Bertilsson M, Holmgren K, Glise K, Pousette A, Segerfelt K, Bjork L. Does employer involvement in primary health care enhance return to work for patients with stress-related mental disorders? a cluster randomized controlled trial. BMC Prim Care. 2023 Sep 20;24(1):195. doi: 10.1186/s12875-023-02151-0. PMID 37730561
- [Derived] Bjork L, Glise K, Pousette A, Bertilsson M, Holmgren K. Involving the employer to enhance return to work among patients with stress-related mental disorders - study protocol of a cluster randomized controlled trial in Swedish primary health care. BMC Public Health. 2018 Jul 6;18(1):838. doi: 10.1186/s12889-018-5714-0. PMID 29976181